CLINICAL TRIAL: NCT02234063
Title: Genomic Medicine Pilot for Hypertension and Kidney Disease in Primary Care
Brief Title: Genetic Testing to Understand and Address Renal Disease Disparities
Acronym: GUARDD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Responsible Party: Principal Investigator, Carol R Horowitz, Professor, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GCO 12-1143
Record Dates: First submitted 2014-09-04; First posted 2014-09-09 (Estimated); Results first posted 2020-10-05 (Actual); Last update posted 2020-10-05 (Actual); Status verified 2020-09

CONDITIONS: Hypertension; Chronic Kidney Disease; Genomics
Keywords: Hypertension; Chronic Kidney Disease; End Stage Renal Disease; APOL1; Genomics; Genetics; Community-engaged
MeSH Terms: conditions — Hypertension; Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Immediate Genetic Testing (Experimental): Participants randomized to intervention will receive the APOL1 genetic test upon study enrollment.
  Interventions: Other: Immediate Genetic Testing
- Control- Delayed Testing (No Intervention): Participants randomized to control will not receive the APOL1 genetic test upon study enrollment. They will be offered the option to take the test during their final follow-up study visit (12 months post enrollment).

INTERVENTIONS:
Other: Immediate Genetic Testing — Participants will receive the APOL1 genetic test. Trained research staff will meet with participants to communicate results and lifetime ESRD risk attributable to variations in the APOL1 gene. Primary care providers will receive APOL1 genetic risk information via a best practice alert in the participant's EMR upon commencement of a patient encounter and through results filed in the participant's genetics results section of their EMR.
  Other Names: Genetic Risk Communication
  Arms: Immediate Genetic Testing

SUMMARY:
In this genomic medicine implementation pilot project, the investigators aim to conduct a randomized trial in a network of community health centers and primary care facilities to study processes, effects and challenges of incorporating information for apolipoprotein L1 (APOL1)-attributable genetic risk for end stage kidney disease in patients of African ancestry with hypertension .

DETAILED DESCRIPTION:
CKD is most commonly associated with diabetes (40%) and hypertension (28%), and affects 26 million American adults. African ancestry populations with hypertension (HTN) have 2- to 3-fold higher risk of developing CKD, and a 5-fold increased risk to progress to end stage renal disease (ESRD) when compared with whites. HTN is a risk factor for progression of CKD and for increased cardiovascular risk with CKD. Thus targeting blood pressure control as a modifiable risk factor may both reduce CVD in people with CKD and reduce progression of CKD to end stage disease. Recent discoveries demonstrate that testable alleles of the APOL1 locus on chromosome 22 have a major effect on and explain almost all of the excess risk for hypertension-associated CKD and its progression to ESRD in African ancestry populations.

We will use community-engaged approaches to enroll patients of African Ancestry with HTN from a network of community health centers and primary care facilities in Harlem and the Bronx and randomize them on a 7 to 1 ratio to receive APOL1 genetic testing and EMR-enabled provider clinical decision support incorporating APOL1 genomic risk information.

ELIGIBILITY:
Inclusion Criteria:

* Ages18-65
* Self-identifies as Black/African American
* History of hypertension
* Patient at a participating site

Exclusion Criteria:

* History of Chronic Kidney Disease
* History of Diabetes
* Pregnant
* Cognitively impaired/unable to provide consent
* Terminally ill
* Planning to leave area of study permanently during the one year study period

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 2052 (Actual)
Dates: Start 2014-11; Primary Completion 2018-01-12 (Actual); Study Completion 2018-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Erwin Bottinger, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai; Carol R Horowitz, MD, MPH, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (2):
- United States (2):
  - Institute for Family Health, New York, New York
  - Icahn School of Medicine at Mount Sinai, New York, New York

REFERENCES:
- [Derived] Nadkarni GN, Fei K, Ramos MA, Hauser D, Bagiella E, Ellis SB, Sanderson S, Scott SA, Sabin T, Madden E, Cooper R, Pollak M, Calman N, Bottinger EP, Horowitz CR. Effects of Testing and Disclosing Ancestry-Specific Genetic Risk for Kidney Failure on Patients and Health Care Professionals: A Randomized Clinical Trial. JAMA Netw Open. 2022 Mar 1;5(3):e221048. doi: 10.1001/jamanetworkopen.2022.1048. PMID 35244702
- See also: Implementing GeNomics In PracTicE (IGNITE) Network Website — https://ignite-genomics.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 15 academic, community and safety-net practices in New York City. 2052 participants were enrolled. however 2 participants were not randomized.
Groups:
- Immediate Genetic Testing: Participants randomized to intervention will receive the APOL1 genetic test immediately upon study enrollment.
Period: Overall Study
Arm/Group | Immediate Genetic Testing | Control- Delayed Testing
Started | 1795 | 255
Completed | 1540 | 212
Not Completed | 255 | 43
Not completed — Lost to Follow-up | 235 | 42
Not completed — Withdrawal by Subject | 20 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control- Delayed Testing | Immediate Genetic Testing | Total
Number analyzed (Participants) | 255 | 1795 | 2050
Age, Continuous [Mean (Standard Deviation); unit: years] | 53 (10) | 53 (10) | 53 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172 | 1187 | 1359
  Male | 83 | 608 | 691
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 255 | 1795 | 2050
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Household income <$30,000/year [Count of Participants; unit: Participants] — Population: Results available for those participants who chose to provide data for this measure.
  Participants
    number analyzed (Participants) | 232 | 1588 | 1820
    (all) | 126 | 888 | 1014
Education more than some college [Count of Participants; unit: Participants] — Population: Results available for those participants who chose to provide data for this measure.
  Participants
    number analyzed (Participants) | 255 | 1791 | 2046
    (all) | 162 | 1008 | 1170
Married/Partner [Count of Participants; unit: Participants] — Population: Results available for those participants who chose to provide data for this measure.
  Participants
    number analyzed (Participants) | 253 | 1791 | 2044
    (all) | 72 | 540 | 612
Type of Insurance [Count of Participants; unit: Participants] — Population: Results available for those participants who chose to provide data for this measure.
  Participants
    Private: number analyzed (Participants) | 255 | 1793 | 2048
    Private | 118 | 745 | 863
    Medicaid | 109 | 821 | 930
    Medicare | 14 | 126 | 140
    Other | 8 | 51 | 59
    None | 6 | 50 | 56
Charlson Comorbidity Index [Count of Participants; unit: Participants] — Charlson Comorbidity Index (CCI) predicts 10-year survival in patients with multiple comorbidities. A score of zero indicates that no comorbidities were found. The higher the score, the more likely the predicted outcome will result in mortality or higher resource use.
  Participants
    0 | 141 | 924 | 1065
    1 | 61 | 481 | 542
    ≥2 | 53 | 390 | 443
Baseline mean Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] — Population: Results available for those participants who chose to provide data for this measure.
  mmHg
    number analyzed (Participants) | 254 | 1795 | 2049
    (all) | 133.8 (19.4) | 134.2 (19.6) | 134.1 (19.5)
Body mass index [Mean (Standard Deviation); unit: kg/m^2] — Population: Results available for those participants who chose to provide data for this measure.
  kg/m^2
    number analyzed (Participants) | 254 | 1795 | 2049
    (all) | 33.9 (7.7) | 32.4 (7.7) | 32.5 (7.6)
Number of Participants with High health literacy [Count of Participants; unit: Participants] — Number of participants who responded with (5) very much confident filling out medical forms.
  Health literacy was assessed at baseline using a single item - "How confident are you filling out medical forms by yourself?" Responses were recorded using a five-point Likert scale of: Not at all confident (1), A little bit confident (2), Somewhat confident (3), Quite a bit confident (4), Very much confident (5). Population: Results available for those participants who chose to provide data for this measure
  Participants
    number analyzed (Participants) | 255 | 1793 | 2048
    (all) | 169 | 1110 | 1279
Excellent/Very good self-reported Health [Count of Participants; unit: Participants] | 64 | 465 | 529

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Urine Protein Excretion
Description: Number of participants with urine protein excretion in urine tests to assess kidney function at 12 months as compared to baseline
Time Frame: Baseline and 12 months
Measure: Count of Participants; unit: Participants
Groups:
- Control- Delayed Testing: Participants randomized to control did not receive the APOL1 genetic test upon study enrollment. They were offered the option to take the test during their final follow-up study visit (12 months post enrollment).
- Immediate Genetic Testing for APOL1 Negative: Participants with low-risk APOL1 alleles (APOL1 negatives) randomized to intervention who received the APOL1 genetic test immediately upon study enrollment.
- Immediate Genetic Testing for APOL1 Positive: Participants with high-risk APOL1 alleles (APOL1 positives) randomized to intervention who received the APOL1 genetic test immediately upon study enrollment.
Arm/Group | Control- Delayed Testing | Immediate Genetic Testing for APOL1 Negative | Immediate Genetic Testing for APOL1 Positive
Number analyzed (Participants) | 255 | 1561 | 234
Participants
  Kidney function urine test before randomization | 33 | 278 | 39
  Kidney function urine test after randomization | 50 | 377 | 68

2. Primary Outcome: Change in Systolic Blood Pressure
Description: Change in systolic blood pressure at 3 months as compared to baseline
Time Frame: Baseline and 3 months
Population: Results available for those participants who returned for 3 month visit and had both timepoint data.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Control- Delayed Testing | Immediate Genetic Testing for APOL1 Negative | Immediate Genetic Testing for APOL1 Positive
Number analyzed (Participants) | 232 | 1468 | 218
mmHg | -3 (18) | -3 (16) | -6 (18)

3. Secondary Outcome: Number of Participants With Change in Medication Adherence
Description: Participant surveys (self-report) regarding medication adherence behaviors 3 months after randomization
Time Frame: 3 months
Population: Survey only for participants who received genetic testing.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Genetic Testing for APOL1 Negative | Immediate Genetic Testing for APOL1 Positive | Control- Delayed Testing
Number analyzed (Participants) | 1468 | 218 | 0
Participants
  Changed how you take BP meds | 146 | 53 |
  Take BP meds more often | 68 | 21 |

4. Secondary Outcome: Number of Patients With Changes in Psychosocial Behaviors
Description: Number of patients with changes in psychosocial behaviors 3 months after randomization
Time Frame: 3 months
Population: Survey only for participants who received genetic testing.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Genetic Testing for APOL1 Negative | Immediate Genetic Testing for APOL1 Positive | Control- Delayed Testing
Number analyzed (Participants) | 1468 | 218 | 0
Participants | 547 | 129 |

5. Secondary Outcome: Number of Participants With Attitude Towards Genetic Testing
Description: Patient attitude towards genetic testing 3 months after randomization
Time Frame: 3 months
Population: Survey only for participants who received genetic testing.
Measure: Count of Participants; unit: Participants
Arm/Group | Immediate Genetic Testing for APOL1 Negative | Immediate Genetic Testing for APOL1 Positive | Control- Delayed Testing
Number analyzed (Participants) | 1468 | 218 | 0
Participants
  Had enough information on getting the test | 1425 | 208 |
  Information for test was easy to understand | 1391 | 203 |
  Would get tested again | 1420 | 211 |

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Control- Delayed Testing | Immediate Genetic Testing for APOL1 Negative | Immediate Genetic Testing for APOL1 Positive
All-Cause Mortality (participants affected / at risk) | 0/255 | 0/1561 | 0/234
Serious Adverse Events (participants affected / at risk) | 0/255 | 0/1561 | 0/234
Other Adverse Events (participants affected / at risk) | 0/255 | 0/1561 | 0/234

LIMITATIONS AND CAVEATS:
Primary analysis was conducted on the Genotype level and not on the randomization level.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-16): https://cdn.clinicaltrials.gov/large-docs/63/NCT02234063/Prot_SAP_000.pdf